CLINICAL TRIAL: NCT01397006
Title: Fibromyalgia of Less Than One Year Duration in Primary Care: Treatment Response in a Double Blind, Placebo Controlled Study of Pregabalin
Brief Title: Fibromyalgia of Less Than One Year Duration. Study of Pregabalin
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Newton-Wellesley Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Don L. Goldenberg MD, PI, Newton-Wellesley Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N11-507
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; pregabalin; Lyrica
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin dose escalating every 2 weeks. Starting dose is 75 mg. Titrated up to maximum of 450mg
  Other Names: Lyrica

SUMMARY:
The purpose of the study is to evaluate whether pregabalin is effective in treating subjects who have had fibromyalgia for less than one year. Pregabalin has been approved by the FDA for treatment of fibromyalgia. the purpose of the study is to see if subjects identified through their primary care physicians who have fibromyalgia and have had symptoms for less than one year respond to pregabalin and to identify characteristics of that response.

DETAILED DESCRIPTION:
The randomized clinical trial of pregabalin in early-onset fibromyalgia.

At the baseline visit, each subject will be asked if they wish to consider enrolling in Part II. If they agree, the details of the study will be explained and Dr Goldenberg will consent those who wish to enroll in Part II. The first 75 patients who consent will be enrolled in the study, the randomized clinical trial of pregabalin in early-onset fibromyalgia.

After a study subject has been enrolled, they will be randomized to one of two treatment groups. All subjects will be randomized, 1:1 either to the pregabalin group (group A) or the placebo group (group B). Randomization will take place after enrollment via selection of one of a multitude of envelopes containing a random number. Each random number will have been preassigned to either Group A or group B.

ELIGIBILITY:
Inclusion Criteria:

* • Meet the 2010 ACR criteria for diagnosis of fibromyalgia (See Appendix)

  * Meet the 1990 ACR criteria for the classification of fibromyalgia (See Appendix)
  * Patients have a pain VAS > 4
  * Patients are able to understand and sign informed consent
  * Patients are able to understand and complete study questionnaires
  * Patients are prepared to discontinue all pain medications including non-steroidal anti-inflammatory drugs (NSAIDs), and medications for sleep or mood disturbances two weeks prior to beginning the study. Acetaminophen, up to 2 extra-strength, three times daily, will be allowed for break-through pain. Medication use will be surveyed at each visit (See Appendix).
  * Age - > 18
  * Females with no documented evidence of current pregnancy, and willingness to take the necessary precautions to prevent pregnancy for the duration of the study period

Exclusion Criteria:

* • Patients with a significant musculoskeletal or rheumatic disorder that may confuse the diagnosis

  * Any subject with suicidal thoughts in the past or currently
  * Patient with a history of renal disease, heart disease, bleeding problems or low platelet counts
  * Women who are breast feeding
  * Men or women who plan to have children during the course of the study
  * Unable to discontinue any medications prescribed for pain, other than acetaminophen, or any medications for sleep or mood disturbances for at least 2 weeks before the study
  * Unable to discontinue any mediations used for sleep disturbances
  * Patients currently being treated for any psychiatric illness including depression or anxiety disorder
  * Patients currently taking antidepressant, anti-anxiety, or antipsychotic medications.
  * Inability to understand and sign informed consent and complete questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in pain VAS from study entry to end of study | 12 weeks

SECONDARY OUTCOMES:
Change in total score FIQ from study entry to last visit. | 12 weeks
Change in total score FM 2010 Clinical Scale from study entry to last visit. | 12 Weeks
Change in PGIC from study entry to last visit. | 12 weeks
Change in total score for HRQOL from study entry to last visit. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Don Goldenberg, MD, Principal Investigator — Newton-Wellesley Hospital
Locations (1):
- Newton-Wellesley Hospital, Newton, Massachusetts, United States

REFERENCES:
- [Background] Goldenberg DL. Fibromyalgia syndrome a decade later: what have we learned? Arch Intern Med. 1999 Apr 26;159(8):777-85. doi: 10.1001/archinte.159.8.777. PMID 10219923
- [Background] Clauw DJ, Crofford LJ. Chronic widespread pain and fibromyalgia: what we know, and what we need to know. Best Pract Res Clin Rheumatol. 2003 Aug;17(4):685-701. doi: 10.1016/s1521-6942(03)00035-4. PMID 12849719
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Goldenberg DL. Introduction: fibromyalgia and its related disorders. J Clin Psychiatry. 2008;69 Suppl 2:4-5. No abstract available. PMID 18537456
- [Background] Goldenberg DL. Pharmacological treatment of fibromyalgia and other chronic musculoskeletal pain. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):499-511. doi: 10.1016/j.berh.2007.02.012. PMID 17602996
- [Result] Goldenberg DL. Fibromyalgia syndrome. An emerging but controversial condition. JAMA. 1987 May 22-29;257(20):2782-7. doi: 10.1001/jama.257.20.2782. PMID 3553636
- [Result] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Result] Crofford LJ, Rowbotham MC, Mease PJ, Russell IJ, Dworkin RH, Corbin AE, Young JP Jr, LaMoreaux LK, Martin SA, Sharma U; Pregabalin 1008-105 Study Group. Pregabalin for the treatment of fibromyalgia syndrome: results of a randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2005 Apr;52(4):1264-73. doi: 10.1002/art.20983. PMID 15818684
- [Result] Mease PJ, Russell IJ, Arnold LM, Florian H, Young JP Jr, Martin SA, Sharma U. A randomized, double-blind, placebo-controlled, phase III trial of pregabalin in the treatment of patients with fibromyalgia. J Rheumatol. 2008 Mar;35(3):502-14. Epub 2008 Feb 15. PMID 18278830
- [Result] Crofford LJ, Mease PJ, Simpson SL, Young JP Jr, Martin SA, Haig GM, Sharma U. Fibromyalgia relapse evaluation and efficacy for durability of meaningful relief (FREEDOM): a 6-month, double-blind, placebo-controlled trial with pregabalin. Pain. 2008 Jun;136(3):419-431. doi: 10.1016/j.pain.2008.02.027. Epub 2008 Apr 8. PMID 18400400
- [Result] Hauser W, Bernardy K, Uceyler N, Sommer C. Treatment of fibromyalgia syndrome with gabapentin and pregabalin--a meta-analysis of randomized controlled trials. Pain. 2009 Sep;145(1-2):69-81. doi: 10.1016/j.pain.2009.05.014. Epub 2009 Jun 17. PMID 19539427